CLINICAL TRIAL: NCT04269278
Title: The Effect of Dexmedetomidine on Blood Coagulation: In Vitro, Volunteer Study Using Rotational Thromboelastometry
Brief Title: Dexmedetomidine and Blood Coagulation
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Associate Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2002/595-301
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Blood Coagulation Disorder
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 0 ng/ml: Blood specimen which was added 0 ul of dexmedetomidine
  Interventions: Drug: 0 ul of dexmedetomidine
- 0.5 ng/ml: Blood specimen which was added 0.25 ul of dexmedetomidine
  Interventions: Drug: 0.25 ul of dexmedetomidine
- 1.0 ng/ml: Blood specimen which was added 0.5 ul of dexmedetomidine
  Interventions: Drug: 0.5 ul of dexmedetomidine
- 1.5 ng/ml: Blood specimen which was added 0.75 ul of dexmedetomidine
  Interventions: Drug: 0.75 ul of dexmedetomidine

INTERVENTIONS:
Drug: 0 ul of dexmedetomidine — Venous blood is taken from 11 healthy volunteers and divided into four specimen bottles, which were added with different doses (0 ul) using dexmedetomidine
  Groups: 0 ng/ml
Drug: 0.25 ul of dexmedetomidine — Venous blood is taken from 11 healthy volunteers and divided into four specimen bottles, which were added with different doses (0.25 ul) using dexmedetomidine
  Groups: 0.5 ng/ml
Drug: 0.5 ul of dexmedetomidine — Venous blood is taken from 11 healthy volunteers and divided into four specimen bottles, which were added with different doses (0.5 ul) using dexmedetomidine
  Groups: 1.0 ng/ml
Drug: 0.75 ul of dexmedetomidine — Venous blood is taken from 11 healthy volunteers and divided into four specimen bottles, which were added with different doses (0.75 ul) using dexmedetomidine
  Groups: 1.5 ng/ml

SUMMARY:
Dexmedetomidine may alter whole blood coagulation. However, little is known about the dose-response relationships according to the blood concentration of dexmedetomidine. The investigators have therefore performed the present study to measure the effect of dexmedetomidine on the coagulation pathway according to the drug concentration level using a rotational thromboelastometry test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age: 20 to 65 years
* Body weight > 50 kg
* Volunteers who provided informed consent

Exclusion Criteria:

* Hematologic disease
* Anticoagulant medication

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
FIBTEM | During the rotational thromboelastometry analysis/ an average of 1 hour
  Fibrinolytic pathway values of rotational thromboelastometry analysis/ FIBTEM is not an acronym.

SECONDARY OUTCOMES:
INTEM | During the rotational thromboelastometry analysis/ an average of 1 hour
  Intrinsic pathway values of rotational thromboelastometry analysis/ INTEM is not an acronym.
EXTEM | During the rotational thromboelastometry analysis/ an average of 1 hour
  Extrinsic pathway values of rotational thromboelastometry analysis/ EXTEM is not an acronym.

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Seok Na, MD., PhD., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Shin HJ, Boo G, Na HS. Effects of dexmedetomidine on blood coagulation: an in vitro study using rotational thromboelastometry. J Anesth. 2021 Oct;35(5):633-637. doi: 10.1007/s00540-021-02969-x. Epub 2021 Jul 15. PMID 34268623